CLINICAL TRIAL: NCT04178811
Title: Holmium Laser Enucleation of Prostate in Management of Benign Prostatic Hyperplasia Patients With Predominant Voiding Versus Storage Lower Urinary Tract Symptoms: A Comparative Retrospective Study
Brief Title: HoLEP in Management of BPH Patients With Predominant Voiding vs Storage LUTS: A Comparative Retrospective Study
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Atef Abdelaziz Mostafa, Assistant Lecturer, Assiut University
Other Study IDs: Benign Prostatic Hyperplasia
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign Prostatic Hyperplasia patients with predominant voiding lower urinary tract symptoms: Outcomes of Holmium Laser Enucleation of Prostate in Management of Benign Prostatic Hyperplasia patients with predominant voiding lower urinary tract symptoms
  Interventions: Device: Holmium Laser Enucleation of Prostate
- Benign Prostatic Hyperplasia patients with predominant storage lower urinary tract symptoms: Outcomes of Holmium Laser Enucleation of Prostate in Management of Benign Prostatic Hyperplasia patients with predominant storage lower urinary tract symptoms
  Interventions: Device: Holmium Laser Enucleation of Prostate

INTERVENTIONS:
Device: Holmium Laser Enucleation of Prostate — Use of Holmium Laser Enucleation of Prostate in management of Benign Prostatic Hyperplasia patients

SUMMARY:
Comparison in outcomes of a minimally invasive surgical modality (Holmium Laser Enucleation of Prostate) in management of voiding versus storage lower urinary tract symptoms associated with Benign Prostatic Hyperplasia

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common condition affecting a large number of men over the age of 50 years and is the major cause of the highly prevalent lower urinary tract symptoms (LUTS) in men of this age group that often necessitate surgical intervention. The LUTS associated with BPH are generally divided into voiding symptoms (slow stream, splitting or spraying, intermittency, hesitancy, straining, terminal dribbling) and storage symptoms (day-time urinary frequency, nocturia, urgency, urinary incontinence). These LUTS are among the most common clinical complaints in adult men with reported increasing prevalence with aging. The storage LUTS may also be termed overactive bladder (OAB) symptoms and are largely encompassed by the term "overactive bladder syndrome" (OABS). While the voiding symptoms are usually more prevalent, the storage symptoms are almost always more bothersome. Associated with a significant burden on both patients and society, these LUTS also have a major impact on patients' quality of life (QoL). As such, The American Urological Association (AUA) has developed the International Prostate Symptom Score (IPSS) as one of the most reliable tools to evaluate the severity of LUTS associated with BPH which, in turn, plays a major role in determining the most appropriate treatment option for BPH.

After being the preferred surgical treatment for BPH patients for more than 30 years, transurethral resection of prostate (TURP) has been replaced by holmium laser enucleation of prostate (HoLEP) as the gold standard surgical treatment for BPH. Introduced in 1995, HoLEP is a minimally invasive surgical procedure that has become the first line treatment of BPH as it provides both effective and safe surgical treatment option for BPH without any size limitation, although at the expense of occasional complications. HoLEP has the advantage of enucleating the enlarging BPH adenoma without destroying the bladder neck thus relieving bladder outflow obstruction (BOO) immediately, safely, and effectively.

Although improvement in both storage and voiding LUTS has been demonstrated after either medical treatment with an alpha-blocker or a 5-alpha-reductase inhibitor or surgical treatment with TURP for BPH patients, few studies have been made to measure the outcomes of HoLEP in BPH-related voiding and/or storage LUTS.

We performed our study with the aim to evaluate and compare the effectiveness and safety of HoLEP in relieving either voiding or storage LUTS in BPH patients.

ELIGIBILITY:
1. Inclusion criteria:

   BPH patients who underwent HoLEP for either predominant voiding or predominant storage LUTS
2. Exclusion criteria:

   1. Active UTI.
   2. PSA ˃ 10 ng/mL (unless negative prostatic biopsy).
   3. Prostatitis within past year.
   4. Previous BPH surgery.
   5. BPH with concomitant bladder stones.
   6. BPH with concomitant neurogenic bladder.
   7. BPH patients with predominant storage LUTS along with PVR of 150 ml or more.
   8. BPH patients taking medications that may mimic or aggravate the LUTS such as antidepressants, diuretics, bronchodilators, anticholinergics, sympathomimetics, and antihistamines (84).
   9. BPH patients having uncontrolled DM or recurrent UTIs.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BPH patients who underwent HoLEP for either predominant voiding or predominant storage LUTS
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | Six months
  Treatment efficacy which will be evaluated by comparing the preoperative urodynamics study (UDS) parameters, patient symptomatology, and international prostate symptom score (IPSS) with their postoperative counterparts.
  International Prostate Symptom Score (IPSS) Minimum Score is Zero. Maximum Score is 35. 0-7 means mildly symptomatic and so good outcome. 8-19 means moderately symptomatic and so worse outcome. 20-35 means severely symptomatic and so worst outcome. Briefly,The lower the score, the better the outcome.

SECONDARY OUTCOMES:
Treatment safety | Six months
  Treatment safety which will be evaluated by collected and analysing any reported complication within the first 6 postoperative months.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Khalil, MD, Study Director — Assiut University; Mohamed A El-Gammal, MD, Study Director — Assiut University; Mohamed A Sayed, MD, Study Director — Assiut University; Ayman Mahdy, MD, Study Chair — University of Cincinnati
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porreca A, D'Agostino D, Vigo M, Corsi P, Romagnoli D, Del Rosso A, Schiavina R, Brunocilla E, Artibani W, Giampaoli M. "In-bore" MRI prostate biopsy is a safe preoperative clinical tool to exclude significant prostate cancer in symptomatic patients with benign prostatic obstruction before transurethral laser enucleation. Arch Ital Urol Androl. 2020 Jan 14;91(4):224-229. doi: 10.4081/aiua.2019.4.224. PMID 31937084
- [Background] Lee YJ, Oh SA, Kim SH, Oh SJ. Patient satisfaction after holmium laser enucleation of the prostate (HoLEP): A prospective cohort study. PLoS One. 2017 Aug 9;12(8):e0182230. doi: 10.1371/journal.pone.0182230. eCollection 2017. PMID 28793314
- [Background] Gratzke C, Schlenker B, Seitz M, Karl A, Hermanek P, Lack N, Stief CG, Reich O. Complications and early postoperative outcome after open prostatectomy in patients with benign prostatic enlargement: results of a prospective multicenter study. J Urol. 2007 Apr;177(4):1419-22. doi: 10.1016/j.juro.2006.11.062. PMID 17382744
- [Background] Martin SA, Haren MT, Marshall VR, Lange K, Wittert GA; Members of the Florey Adelaide Male Ageing Study. Prevalence and factors associated with uncomplicated storage and voiding lower urinary tract symptoms in community-dwelling Australian men. World J Urol. 2011 Apr;29(2):179-84. doi: 10.1007/s00345-010-0605-8. Epub 2010 Oct 21. PMID 20963421
- [Background] Saito K, Hisasue S, Ide H, Aoki H, Muto S, Yamaguchi R, Tsujimura A, Horie S. The Impact of Increased Bladder Blood Flow on Storage Symptoms after Holmium Laser Enucleation of the Prostate. PLoS One. 2015 Jun 19;10(6):e0129111. doi: 10.1371/journal.pone.0129111. eCollection 2015. PMID 26090819
- [Background] Peters TJ, Donovan JL, Kay HE, Abrams P, de la Rosette JJ, Porru D, Thuroff JW. The International Continence Society "Benign Prostatic Hyperplasia" Study: the botherosomeness of urinary symptoms. J Urol. 1997 Mar;157(3):885-9. PMID 9072592
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Rodrigues P, Meller A, Campagnari JC, Alcantara D, D'Imperio M. International Prostate Symptom Score--IPSS-AUA as discriminat scale in 400 male patients with lower urinary tract symptoms (LUTS). Int Braz J Urol. 2004 Mar-Apr;30(2):135-41. doi: 10.1590/s1677-55382004000200011. PMID 15703098
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] O'Leary MP, Wei JT, Roehrborn CG, Miner M; BPH Registry and Patient Survey Steering Committee. Correlation of the International Prostate Symptom Score bother question with the Benign Prostatic Hyperplasia Impact Index in a clinical practice setting. BJU Int. 2008 Jun;101(12):1531-5. doi: 10.1111/j.1464-410X.2008.07574.x. Epub 2008 Apr 28. PMID 18445080
- [Background] Jeong J, Lee HS, Cho WJ, Jung W, You HW, Kim TH, Sung HH, Lee KS. Effect of Detrusor Overactivity on Functional Outcomes After Holmium Laser Enucleation of the Prostate in Patients With Benign Prostatic Obstruction. Urology. 2015 Jul;86(1):133-8. doi: 10.1016/j.urology.2015.03.033. Epub 2015 May 16. PMID 25991576